CLINICAL TRIAL: NCT06519110
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Study of Neratinib Tablets Monotherapy in the Treatment of Advanced Solid Tumors With HER2 Mutations
Brief Title: Neratinib Tablets Monotherapy for Advanced Solid Tumors With HER2 Mutations
Acronym: CVL009-C2001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL009-C2001
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor
Keywords: HER2 mutation-positive; Non-Small Cell Lung Cancer (NSCLC); Cholangiocarcinoma; Cervical Cancer; Salivary Gland Cancer; Neratinib tablets
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Uterine Cervical Neoplasms; Salivary Gland Neoplasms | interventions — neratinib

STUDY DESIGN:
Intervention Model Description: Patients with advanced solid tumors (non-small cell lung cancer, cholangiocarcinoma, cervical cancer, salivary gland cancer) with HER2 mutations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (Trial group)-Neratinib tablets (Experimental): The subjects enrolled in the study will take Neratinib tablets orally as follows: 120mg in the 1st week, 160mg in the 2nd week, and 240mg from the 3rd week until the end of treatment (starting from C1D15 to the end of treatment). During the Neratinib treatment period, loperamide will be administered on an as-needed basis based on the condition of diarrhea.
  Neratinib tablets should be taken orally once daily, with the tablet to be swallowed whole with a meal, without crushing, breaking, or chewing. A continuous 28-day medication period constitutes one treatment cycle.
  Interventions: Drug: Neratinib tablets

INTERVENTIONS:
Drug: Neratinib tablets — In the first week, take Neratinib tablets 120mg orally, in the second week take Neratinib tablets 160mg orally, and from the third week until the end of treatment, take Nilotinib tablets 240mg orally (from Cycle 1 Day 15 until the end of treatment).
  Other Names: Neratinib

SUMMARY:
Evaluating the efficacy of Neratinib tablets monotherapy in treating advanced solid tumors with HER2 mutations.

DETAILED DESCRIPTION:
This single-arm, open-label, multicenter Phase II clinical study is divided into three phases: screening, treatment, and follow-up. The screening phase occurs within 28 days prior to the first administration of the study drug. During the treatment phase, a 28-day cycle is used, and tumor efficacy is assessed according to the RECIST 1.1 criteria. Assessments are conducted at the end of the first cycle (±3 days), followed by imaging evaluations every 8 weeks until disease progression. During the treatment period, the investigator may increase the number of assessments based on clinical needs. The study drug will be administered continuously until intolerable adverse reactions occur, disease progression, withdrawal of informed consent, loss to follow-up, death, or study termination.

The follow-up phase includes safety and survival follow-up. Safety follow-up occurs within 28 days after the last administration of the study drug. Survival follow-up is conducted every 12 weeks to collect the survival status of the subjects until their death, loss to follow-up, withdrawal from the study, or study termination (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* 1.Age is 18 years or older, and the patient can be male or female;
* 2.Histologically or cytologically confirmed advanced non-small cell lung cancer, cholangiocarcinoma, cervical cancer, and salivary gland cancer patients; those who have failed to respond to ≤2 lines of standard treatment (disease progression after treatment or intolerable toxic side effects of treatment), or have no standard treatment options, or are unable to receive standard treatment;
* 3.Previously underwent second-generation sequencing testing with evidence of HER2 mutation, otherwise, the patient must provide sufficient tissue samples for second-generation sequencing testing in the study's central laboratory, with tissue samples being the primary source; if tissue slices or samples that meet the requirements cannot be obtained, blood samples may be provided for testing.
* 4.According to the RECIST v1.1 criteria (see Appendix 1), there must be at least one measurable lesion; if the only lesion is one that has previously received local treatment (such as radiotherapy, ablation, interventional treatment, etc.), there must be clear radiological evidence of disease progression;
* 5.Eastern Cooperative Oncology Group (ECOG) performance status score is 0-1;
* 6.Predicted survival is 3 months or more;
* 7.Bone marrow reserve must meet the following laboratory value criteria: Absolute neutrophil count (ANC) is ≥1.5 × 10^9/L; Platelet count (PLT) is ≥90 × 10^9/L; Hemoglobin (Hb) is ≥90 g/L; Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) are ≤2.5 × ULN (the upper limit of the normal range); if liver metastasis is present, it should be ≤5 × ULN; Total bilirubin (TBIL) is ≤1.5 × ULN; Blood urea/urea nitrogen (UREA/BUN) and Creatinine (Cr) are ≤1.5 × ULN; Coagulation function: International normalized ratio (INR) and Activated partial thromboplastin time (APTT) are ≤1.5 × ULN; Urine protein is less than 2+ (if baseline urine protein is ≥2+, a 24-hour urine protein quantification should be performed, and it is acceptable for inclusion if ≤1g);
* 8.Women of reproductive age should agree to use contraceptive measures (such as intrauterine devices, hormonal contraceptives, or condoms) during the study period and for 6 months after the study ends; they must have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must not be breastfeeding; men should agree to use contraceptive measures during the study period and for 6 months after the study ends;
* 9.The subject can understand the nature of this study, and the subject and/or legal representative voluntarily agrees to participate in this trial and signs the informed consent.

Exclusion Criteria:

* 1.Patients who have previously received treatment with any HER2-targeted tyrosine kinase inhibitors (such as lapatinib, pyrotinib, neratinib, etc.);
* 2.Those who do not meet the following requirements for the washout period from previous anti-tumor treatments before the first administration of the study drug: the washout time from the end of the last dose of previous anti-tumor treatment to the first administration of the study drug (calculated from the end of the last dose) is as follows: chemotherapy ≥3 weeks (oral fluorouracil ≥2 weeks; mitomycin C, nitrosoureas ≥6 weeks), small molecule targeted therapy ≥2 weeks, large molecule drugs (including immunotherapy) ≥4 weeks, radiotherapy ≥4 weeks (local palliative radiotherapy ≥2 weeks), Chinese medicine with anti-tumor indications ≥2 weeks, other anti-tumor treatments ≥4 weeks, investigational drugs or treatments that are not yet marketed ≥4 weeks;
* 3.Received major organ surgery (excluding biopsy) or had significant trauma within 4 weeks before the first administration of the study drug;
* 4.Spinal cord compression or brain metastasis, unless asymptomatic, stable, and has not required steroid treatment for at least 4 weeks before the start of the study treatment (before dosing);
* 5.A history of other malignant tumors within the past 5 years, excluding cured cancers such as cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin;
* 6.Adverse reactions from previous anti-tumor treatments have not recovered to a grade of ≤1 according to CTCAE 5.0 (except for toxicities judged by the investigator to have no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, thyroid hypothyroidism stable with hormone replacement therapy);
* 7.The presence of uncontrollable third-space fluid accumulation (such as a large amount of pleural effusion, ascites, or pericardial effusion) that cannot be managed by drainage or other methods;
* 8.Patients with gastrointestinal diseases that may affect drug absorption (such as Crohn's disease, intestinal obstruction, active peptic ulcer disease, etc.);
* 9.Patients currently suffering from interstitial lung disease;
* 10.Patients with any cardiac disease, including: (1) unstable angina; (2) clinically significant arrhythmias requiring medication; (3) myocardial infarction; (4) heart failure of grade 3 or higher; (5) echocardiography: left ventricular ejection fraction (LVEF) ≤50%; (6) 12-lead electrocardiogram: QTcF: females >470 milliseconds, males >450 milliseconds; (7) any other cardiac disease judged by the investigator to be unsuitable for participating in this trial;
* 11.History of immunodeficiency, including HIV antibody test positive;
* 12.Active hepatitis B or C (HBV DNA, HCV RNA test results at screening are not within the normal range of the central laboratory);
* 13.According to the investigator's judgment, there are other serious accompanying diseases that endanger patient safety or affect the patient's ability to complete the study (such as uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg after taking antihypertensive drugs), diabetes (glycated hemoglobin >9.0%), autoimmune diseases, etc.);
* 14.The investigator deems the subject unsuitable for other reasons to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rates of the central nervous system as assessed by the Independent Imaging Evaluation Committee based on RECIST1.1 | Throughout the study for approximately 3.5 years
  Objective response rates of the central nervous system as assessed by the Independent Imaging Evaluation Committee based on RECIST1.1

SECONDARY OUTCOMES:
Duration of Response (DoR) | Throughout the study for approximately 3.5 years
  DoR as assessed by the investigator
Progression-Free Survival (PFS) | Throughout the study for approximately 3.5 years
  PFS as assessed by the investigator
Disease Control Rate (DCR) | Throughout the study for approximately 3.5 years
  DCR as assessed by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: jin Li, ph.D, Principal Investigator — Shanghai GoBroad Cancer Hospital China Pharmaceutical University

IPD SHARING:
Plan to Share IPD: No